CLINICAL TRIAL: NCT01358669
Title: Effect of Denosumab on Inflammatory Osteolytic Lesion Activity in Total Hip
Brief Title: Effect of Denosumab on Inflammatory Osteolytic Lesion Activity in Total Hip Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Amgen (Industry); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STH15714
Record Dates: First submitted 2011-05-11; First posted 2011-05-24 (Estimated); Last update posted 2022-08-29 (Actual); Status verified 2019-11

CONDITIONS: Revision Surgery of Total Hip Arthroplasty
Keywords: Denosumab; Total Hip Arthroplasty
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab (Active Comparator): In this study we explore the potential for giving a medication (denosumab) that may prevent the loss of bone around the hip replacement implant
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Denosumab — 60mg denosumab by injection as a single dose
  Other Names: Prolia
  Arms: Denosumab
Other: Placebo — Placebo by injection as a single dose
  Arms: Placebo

SUMMARY:
Although hip replacement surgery is a successful way of dealing with the pain and immobility caused by hip arthritis, 10% of the hip replacements carried out in the UK fail within 10 years. The main reason for this is the development periprosthetic osteolysis, that is, loss of bone around the site of the hip replacement. The osteolysis is thought to be due to the small particles of debris worn from the surfaces of the hip implant. These particles cause a reaction in the blood cells around the joint which in turn affects bone cells and leads to a loss of bone around the implant. The joint implant will then eventually become loose and unstable, a condition known as aseptic loosening. At present the only way to treat aseptic loosening is to have another operation to secure the hip joint, known as revision surgery. Revision surgery is not always successful and exposes the patient to the risk of major surgery.

In this study we explore the potential for giving a medication (denosumab) that may prevent the loss of bone around the hip replacement implant. We will recruit patients who have been listed for revision surgery. One group of patients will be given a single dose of denosumab; another group will be given a placebo (dummy drug). At the time of the revision surgery a small sample of the bone from around the hip replacement will be taken and examined under the microscope. Comparisons will be made between the patients having the denosumab and those having placebo to find out whether the denosumab is having a beneficial effect on the bone surfaces. If successful, this study will lead to further studies to develop the use of denosumab to prevent aseptic loosening.

DETAILED DESCRIPTION:
This is a single centre, double blinded, randomized, controlled trial of denosumab compared to placebo in adults undergoing revision surgery of total hip arthroplasty due to prosthesis related osteolysis. A total of 30 subjects will be enrolled into the study. Subjects will be randomized to receive either denosumab or placebo. 15 participants will be assigned to each treatment arm.

1. 60mg denosumab by injection as a single dose
2. Placebo by injection as a single dose After they have given informed consent, all participants will have a screening visit (Visit 1). Participants who are eligible after completing all screening assessments will be randomly assigned to receive one of the two treatments. All screening procedures will be completed within 14 (±7) days before beginning the medication. Study medication will be given at visit 2, which will occur 8 weeks (56 ±7 days) before the date of the planned revision surgery. Participants will attend for 5 visits in total as shown below. Visit 1, Baseline, 2 weeks (±7 days)before being given the study medication

   * Informed consent
   * Personal and demographic data
   * Medical history
   * Physical exam
   * Weight and height
   * Concomitant medication (other medications being taken at the visit)
   * Blood samples for eligibility, and bone turnover markers
   * Urine samples for bone turnover markers
   * Vital signs including blood pressure (BP), heart rate (HR) and temperature
   * Personal and demographic data
   * Medical history
   * Physical exam
   * Weight and height
   * Concomitant medication (other medications being taken at the visit)
   * Blood samples for eligibility, and bone turnover markers
   * Urine samples for bone turnover markers
   * Vital signs including blood pressure (BP), heart rate (HR) and temperature Visit 2, Randomization and administration of denosumab or placebo (day 0)
   * Blood sampling for bone turnover markers
   * Urine sampling for bone turnover markers
   * Changes to medical history
   * Changes to concomitant medications
   * Record of adverse events
   * Oxford and Harris hip scores (by questionnaire)
   * Pregnancy test if applicable
   * Administration of medication
   * Vital signs including BP, HR and temperature
   * Conebeam CT scan of the affected hip Visit 3, Week 4 (±7 days)
   * Blood sampling for bone turnover markers
   * Urine sampling for bone turnover markers
   * Changes to medical history
   * Record of adverse events
   * Record of concomitant medications
   * Oxford and Harris hip scores
   * Vital signs including BP,HR and temperature
   * Check on injection site Visit 4, Week 8 (±14 days) (Revision Surgery)
   * Standard preoperative admission procedures
   * Blood sampling for bone turnover markers
   * Urine sampling for bone turnover markers
   * Changes to medical history
   * Adverse events recorded
   * Record of concomitant medications
   * Oxford and Harris hip scores
   * Bone and tissue biopsy
   * Vital signs including BP, heart rate and temperature Visit 5, Week 14 (±7 days) (Safety follow up visit)
   * Blood sampling for bone turnover markers
   * Urine sampling for bone turnover markers
   * Changes to medical history
   * Adverse events recorded
   * Record of concomitant medications
   * Oxford and Harris hip score
   * Vital signs including BP and heart rate
   * Pregnancy test if applicable
   * Plain Xray of the pelvis and hip

ELIGIBILITY:
Inclusion Criteria:

* Participants must be men or women over 30 years of age undergoing revision THA surgery for periprosthetic osteolysis / aseptic loosening affecting the pelvis and / or femur.
* Participants must also be willing and able to give fully informed consent.
* Participants must have osteolysis / aseptic loosening affecting fully cementless, hybrid, or fully cemented THA prosthesis

Exclusion Criteria:

* Known prosthesis infection
* Pregnancy / Breast feeding
* Oral bisphosphonate therapy (current use, previous use within the last 12 months, previous 3 or more years cumulative use)
* Administration of intravenous bisphosphonate, fluoride or strontium within the last 5 years
* Participation in ongoing or previous denosumab clinical trials
* Administration of any of the following treatments within the last 12 months
* TH or PTH derivatives, eg, teriparatide
* anabolic steroids or testosterone
* glucocorticosteroids (> 5 mg prednisone equivalent per day for more than 10 days)
* systemic hormone replacement therapy
* selective estrogen receptor modulators (SERMs), eg, raloxifene tibolone, calcitonin or calcitriol
* Any subject in whom denosumab is contraindicated according to the local SmPC of denosumab (SC 60 mg every 6 months in UK)
* Current hypocalcemia (albumin adjusted serum calcium below 2.13 mmol/L)
* History of rheumatoid arthritis
* History of Paget's disease
* Malignancy (except basal cell carcinoma, cervical or breast ductal carcinoma in situ) within the last 5 years
* Renal insufficiency assessed by eGFR <30
* Known sensitivity to mammalian cell derived drug products
* Any organic or psychiatric disorder, or laboratory abnormality which, in the opinion of the Investigator, will prevent the subject from completing the study or interfere with the interpretation of the study results
* Any disorder that, in the opinion of the Investigator, may compromise the ability of the subject to give written informed consent and/or comply with study procedures
* Evidence of alcohol or substance abuse within the last 12 months that the Investigator believes would interfere with understanding or completing the study
* Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12-14 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Osteoclast number | 8 weeks after administration
  Absolute difference between study groups in osteoclast number per millimetre at the osteolysis membranebone interface, measured by cell counting in histological sections between the denosumab and placebo groups, 8 weeks after administration of the IMP

SECONDARY OUTCOMES:
Change in serum or urine levels of βCTXI, NTXI/Cr, TRAcP5b, CTXMMP, PINP, OPG, RANKL | 8 weeks after administration of the IMP
  Difference between the denosumab and placebo groups in mean absolute change in serum or urine levels of βCTXI, NTXI/Cr, TRAcP5b, CTXMMP, PINP, OPG, RANKL, 8 weeks after administration of the IMP
Difference between the denosumab and placebo groups in mean eroded, quiescent, and osteoblast surfaces at the membrane bone interface | 8 weeks after administration of the IMP
  Difference between the denosumab and placebo groups in mean eroded, quiescent, and osteoblast surfaces at the membrane bone interface measured using image analysis software, 8 weeks after administration of the IMP (Bioquant Image Analysis Corp, Nashville, TN, USA)
Difference between the denosumab and placebo groups in ratio of viable to apoptotic osteoclast, macrophage fibroblast, and osteoblasts by TUNEL staining and relative number of cells staining positive for apoptosis markers | 8 weeks after administration of the IMP
  Difference between the denosumab and placebo groups in ratio of viable to apoptotic osteoclast, macrophage fibroblast, and osteoblasts by TUNEL staining and relative number of cells staining positive for apoptosis markers, including but not limited to, Caspase 8, 9, and 3, and proliferation marker Ki67 8 weeks after administration of the IMP

CONTACTS AND LOCATIONS:
Overall Officials: J M Wilkinson, PhD, FRCS (Tr&Orth), Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust/University of Sheffield
Locations (1):
- Academic Unit of Bone Metabolism, Sheffield, South Yorkshire, United Kingdom